CLINICAL TRIAL: NCT03493906
Title: Patient Ambassador Support in Newly Diagnosed Patients With Acute Leukemia During Treatment: a Feasibility Study
Brief Title: Patient Ambassador Support in Newly Diagnosed Patients With Acute Leukemia During Treatment
Acronym: PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristina Holmegaard Nørskov, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Rigshospitalet PAS
Record Dates: First submitted 2018-01-05; First posted 2018-04-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patient Ambassador Support
  Interventions: Other: Patient Ambassador Support

INTERVENTIONS:
Other: Patient Ambassador Support — Patient Ambassador Support, with former patient treated for acute leukaemia being ambassadors for newly diagnosed patients for a period of 12 weeks.

SUMMARY:
Background: Acute leukemia is a life threatening hematological malignancy which can result in substantial symptom burden including impaired psychological wellbeing. Peer-to-peer support has positive and beneficial effects on patients with cancer. Yet there is lack of knowledge and evidence of the feasibility and the effect of peer-to-peer support on patient with acute leukemia

Aims: The study aim to examine the feasibility and safety of Patient Ambassador Support in newly diagnosed patients with acute leukemia during treatment, and to examine the benefit on symptoms and psychological wellbeing in both patients and ambassadors.

Design and methods: This study is a one arm feasibility intervention trial with patients n=40; patient ambassadors (PA) n=30. Patients will be consecutively recruited at the Departments of Hematology, Rigshospitalet, Herlev and Gentofte Hospital and Sjællands Universitetshospital, Roskilde, and paired with a PA who will follow and assist the patient over the course of two series of chemotherapy for a 12 week period, with one follow-up contact at 3 month. Data is collected at baseline (within 2 weeks of diagnosis), post intervention (12 weeks) and follow-up 6 months.

Implication: This study has the potential to be a new model for care incorporated in the oncology/hematology clinical care setting, creating an active partnership between patients and former patients; and in collaboration with the health care professionals which may strengthen the existing care and support system.

DETAILED DESCRIPTION:
Study Part 2 Aim To investigate the feasibility and safety of Patient Ambassador Support (PAS) and whether there is benefit on psychological wellbeing and symptoms among newly diagnosed patients with acute leukemia and among former patients with acute leukemia (patient ambassadors).

Design and Methods A one arm feasibility intervention trial with patients (n=40) and patient ambassadors (PA) (n=30).

Recruitment Patients will be recruited at three Danish hematology departments: Rigshospitalet (RH), Herlev og Gentofte Hospital (HGH and Sjællands Universitetshospital, Roskilde (SUR), from January 2018 to June 2019. Eligible patients receive oral and written project information from KHN within two weeks from diagnosis. KHN provides a summary of the study and gives the opportunity to raise questions or concerns related to the study.

PA´s will be recruited voluntarily from the patient association LyLe and from the outpatient hematology departments of RH, HGH and SUR by KHN, and screened by interview to assess their appropriateness for the intervention. Screening interviews include questions about a survivor´s motivation for volunteering, availability, ability to respect confidentiality, and ability to acknowledge the vulnerability that may occur when they revisiting experience of others with acute leukemia. The PA is obligated to sign a confidentiality commitment, and knows and accepts the terms and requirements included in the intervention. Furthermore, the PA provides information regarding age, gender, diagnose, treatment, interests, work, education, social conditions in order to match with patients. The PA must provide transportation themselves but will receive a monetary incentive for their participation. During the intervention we will adjust the PA recruitment process in order to fill specific needs in the program such as age groups or diagnosis. This will ensure that we do not have a larger ambassador pool than we effectively utilize.

Patients and ambassadors who have consented and agreed to participate in the study will complete the baseline testing (patient reported outcome questionnaires) before the beginning of intervention.

Patient ambassador training program Recruited PAs will receive a group training program, curriculum and an ambassador 'checklist´. Before interacting with patients, the PA will receive 6 hours of training. The training will be organized by KHN and a project nurse from each intervention site. The training will be carried out by KHN, the project nurse, a represent from the PAB and a psychologist. Training modules include information on medical facts related to acute leukemia, information on psychosocial issues, training in communication skills with emphasis on active listening, and learning how to help other patients problem- solve and advocate for themselves within the health care system. Training also includes discussion of the PA ´s personal goals and concerns about volunteering in the study and their individual attitudes toward survivorship and illness. The importance of maintaining appropriate boundaries are discussed, to ensure PA do not overly identify with patients and remain aware of their role as listening mentors who use their experience only when solicited by the patient. Further, possible changes in medical conditions in both themselves and the patients will be discussed. The PA is offered supervision during the intervention and the opportunity to attend ambassador support meetings every second month for ongoing education and to process their experiences with patients.

Match between patients and ambassadors Patients and ambassadors express prior to intervention which preferences they have for their match. They will be matched according to diagnosis, age, gender and other factors that might create a mutual understanding and ease of communication. KHN will pair patients with a PA. If it is not possible to match on the given preferences, the patient and ambassador will be involved in the decision.

PAS intervention The intervention consists of support provided by the PA, who will follow and assist the patient over the course of 12 weeks, through two series of chemotherapy. The intervention consists of minimum four face-to-face meetings between patient and PA and additionally open telephone and/or email contact based on the patients 'individual needs, including one follow-up contact at 3 months by telephone. The duration of the contact is individual. The context of the face-to-face meetings are chosen between patients and ambassadors e.g. café on the local hospital, a café near both patient and ambassador or private based on the contact developed between patient and ambassador. The PA will follow one patient at a time, however at the end of the 12 week period; the PA can choose to follow a new patient. During the first meeting, an expectation agreement between the patient and PA will be discussed and signed. The PA will use an ambassador checklist to document the frequency, content and quality of the connections between patient and PA, as well as documenting themes, goals, progress and outcomes of their conversations. The checklist will be developed in conjunction with representatives from the PAB and prior to the recruitment of the IG. The checklist will provide a comprehensive guidance and list of important and relevant actions, or steps to be taken in the role as PA, as well as serve as a work and documentation tool during the intervention and follow-period. Upon completion of the training program each PA will receive a training certificate and a personal PA name badge.

Changes in medical conditions in both patients and ambassadors which will affect their ability to participate in the study will result in exclusion. The project nurse at the specific hematologic department reports to the primary investigator (KHN) within 48 hours. Changes in medical conditions comprise the following conditions: relapse (ambassadors), critical psychological conditions including delirium or severe depression, hospitalization in intensive care unit (ICU) longer than two weeks or transition to palliative care.

Safety net - ambassadors' support There will be held an ambassador support meeting which is important to allow the ambassadors to share experiences, solve problems, and provide mutual support. The ambassadors have the possibility to request supervision from a psychologist during the intervention. The psychological health of the ambassadors is of great interest and it is important that they do not suffer unnecessary distress following the intervention. Any adverse events will be documented and acted on.

Outcomes measurements and data collection Data are collected by patient reported outcome measures (PROM) completed by patients electronically prior to intervention, post intervention (12 weeks) and at 3-month follow-up. PROM is completed by PA, after they have completed the patient ambassador training program, but prior to their first PAS intervention and at post intervention (12 weeks). Socio-demographic characteristics are collected through by patient's medical charts and questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are > 18 years and newly diagnosed with acute leukemia < 2 weeks of diagnosis who are planned to receive intensive treatment during a course of minimum two series of chemotherapy, and ambassadors (PA) > 18 years who have completed treatment for their acute leukemia > 6 month (in complete remission) and provides consent to participate in the ambassador training program, and applicable to all participants (patients and PA) written informed consent is provided.

Exclusion Criteria:

* Patients and ambassadors are excluded if they do not understand, read and speak Danish, if they have unstable medical disease or cognitive / psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 2 years
  Number of participants included from eligible patients
Adherence to intervention | Up to 24 weeks
  number of weeks completed out of planned weeks of intervention
Emotional reactions (Total numbers of contacts with project team members) | Up to 24 weeks
  Measured by registration on numbers of contact made by participants to primary investigator / project psychologist / project nurse
Emotional reactions (content of contacts with project team members) | Up to 24 weeks
  Measured by registration quality of contact made by participants to primary investigator / project psychologist / project nurse

SECONDARY OUTCOMES:
Quality Of Life | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the EORTC Quality of Life Questionnaire (EORTC QLQ-C30)
Symptom burden | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the M.D. Anderson Symptom Inventory (MDSAI) patient questionnaire
Patient Activation Measure | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the Patient activation measure (PAM) questionnaire
Anxiety and Depression | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the The Hospital Anxiety and Depression Scale (HADS) patient questionnaire
Quality of Life | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the Functional Assessment of Cancer Therapy - Leukemia (FACT-LEU)
Self-efficacy | Change measures (baseline, 12 weeks, and 24 weeks)
  Measured with the The General Self-Efficacy Scale patient questionnaire
Hospital admissions (total number of admissions) | Up to 24 weeks
  Data will be collected from medical charts
Hospital admissions (causes) | Up to 24 weeks
  Data will be collected from medical charts
Hospital admissions (days) | Up to 24 weeks
  Data will be collected from medical charts
Proportion of participants with overall survival up to 24 weeks | Up to 24 weeks
  Data will be collected from medical charts
Infections (type) | Up to 24 weeks
  Data will be collected from medical charts
Infections (days) | Up to 24 weeks
  Data will be collected from medical charts
Physical activity level | Change measures (baseline, 12 weeks, and 24 weeks)
  Leisure Time Physical Activity Scale
Number of contacts between patient and ambassador | Up to 12 weeks
  Measured by the total number of contacts during 12 week of intervention
Length of contacts between patient and ambassador | Up to 12 weeks
  Measured by the total time of contacts during 12 week of intervention
Thematic content of the contacts between patient and ambassador | Up to 12 weeks
  Measured by ambassadors thematic registration of the contacts with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Jarden, ph.d., Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Herlev Hospital, Herlev
  - Sjællandsuniversitetshospital Roskilde, Roskilde
  - Rigshospitalet, Copenhagen, Østerbro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noerskov KH, Nielsen IH, Rahbaek ES, Halbro S, Mortensen AO, Overgaard UM, Piil K, Jarden M. Implementation and Evaluation of Peer Ambassador Support to Patients Newly Diagnosed With Hematological Cancer and Their Caregivers. Nurs Res Pract. 2025 Apr 28;2025:4528051. doi: 10.1155/nrp/4528051. eCollection 2025. PMID 40330711
- [Derived] Norskov KH, Overgaard D, Boesen J, Struer A, El-Azem SEWD, Tolver A, Lomborg K, Kjeldsen L, Jarden M. Patient ambassador support in newly diagnosed patients with acute leukemia during treatment: a feasibility study. Support Care Cancer. 2021 Jun;29(6):3077-3089. doi: 10.1007/s00520-020-05819-w. Epub 2020 Oct 13. PMID 33051828